CLINICAL TRIAL: NCT00597142
Title: A Prospective, Multi-center, Single Arm Study Evaluating the Express™ Renal Premounted Stent System in the Treatment of Atherosclerotic Lesions in the Aortorenal Ostium.
Acronym: RENAISSANCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2006
Record Dates: First submitted 2008-01-09; First posted 2008-01-17 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Atherosclerotic Lesions in the Aortorenal Ostium
Keywords: renal stent; stent; atherosclerosis; aortorenal ostium; renal; renal artery; PTRA
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Express™ Renal Premounted Stent System

INTERVENTIONS:
Device: Express™ Renal Premounted Stent System — This device is indicated for use as an adjunct to percutaneous transluminal renal angioplasty (PTRA) of a:
  * Single, de novo or restenotic (from PTRA) atherosclerotic lesion in the ostium of the renal artery
  * Lesion length ≤15mm
  * Lesion involving the aortorenal ostium or the leading edge of the stenosis is located within 5 mm of the opacified aortic lumen
  * RVD 4.0-7.0mm

SUMMARY:
The purpose of this study is to demonstrate superior 9-month binary restenosis rate of the Express™ Renal Premounted Stent System as compared to an Objective Performance Criterion representative of PTRA, for atherosclerotic lesions in the aortorenal ostium.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for PTRA and stenting.
* One or more of the following: (1-3)
* Hypertension
* Recurrent "flash" pulmonary edema out of proportion to any impairment of left ventricular function
* Renal Dysfunction
* Single, de novo, or restenotic (from prior PTRA) atherosclerotic lesion in the ostium of the renal artery
* Lesion involving the aortorenal ostium or the leading edge of the stenosis is located within 5 mm of the opacified aortic lumen
* Renal Artery Stenosis: bilateral renal artery stenosis (one stent for one lesion in each renal artery) or unilateral renal artery stenosis, including a solitary functioning kidney

Exclusion Criteria:

* Any previous or planned, surgery or percutaneous intervention ≤30 days prior to or after index procedure
* Advanced renal disease: serum creatinine > 3.0 mg/dl
* End stage renal disease requiring dialysis; or previously diagnosed ephrosclerosis
* Recent vascular event ≤30 days pre-procedure (i.e. acute coronary syndrome, decompensated heart failure, transient ischemic attack or stroke.)
* Documented allergy or reaction to iodinated contrast media, including laryngeal edema, convulsions, profound hypotension,unresponsiveness, cardiopulmonary arrest, and clinically manifest arrhythmias (a mild allergy to contrast media that can be pretreated with medication is acceptable)
* Documented allergy to heparin, acetylsalicylic acid (ASA) or clopidogrel
* NYHA Class IV
* Bleeding diathesis
* Thrombocytopenia (platelets < 100,000/mm3)
* Renal atrophy (renal length ≤ 8 cm determined by renal ultrasound)
* Patients requiring immunosuppressive therapy
* Renal allograft
* Stenosis location in a vascular graft or in a transplant artery Angiographic Exclusion
* Total occlusions
* Thrombus containing lesion
* Prior treatment of target lesion with stent (in-stent restenosis)
* More than one (1) lesion in target vessel
* Non-atherosclerotic stenosis (fibromuscular dysplasia)
* Excessive vessel tortuosity
* Lesion involving a side-branch
* Lesion in accessory renal artery
* Abdominal aortic aneurysm > 3.5 cm
* Perforated vessels evidenced by extravasation of contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-01; Primary Completion 2005-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Binary in-stent restenosis rate of the Express™ Renal Stent at nine (9) months, defined by quantitative angiography. | 9 months

SECONDARY OUTCOMES:
Procedural Success - <30% residual diameter stenosis as visually assessed by the investigator without the occurrence of in-hospital MAE. | Post stent deployment
Target Lesion Revascularization(TLR)*- Clinically driven reintervention of the target lesion through 9-months. | 9 months
Target Vessel Revascularization(TVR)* - Clinically driven reintervention of the target vessel through 9-months. | 9 Months
Change (improvement) in renal function from pre-procedure to post-procedure, 1-month and 9-month followups | 9 months
Change in Renal to Aortic Ratio, Resistive Index, and Peak Systolic Velocity using Ultrasound Core Lab values from pre-procedure to postprocedure and 9-months post-procedure. | 9 Months
Change (improvement) in hypertension control from pre-procedure to post-procedure, 30-day and 9-month followups | 9 Months
Major Adverse Events (MAEs): device- or index procedure related death ,TLR, Significant Embolic Event through 9 months post-procedure | 9 Months
Technical success as visually assessed by the investigator. | Immediately after stent deployment

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Grady, PhD, Study Director — Boston Scientific Corporation; Krishna Rocha-Singh, MD, Principal Investigator — Prairie Cardiovascular Heart Institute, St. John's Hospital
Locations (14):
- United States (14):
  - Sarasota Memorial Hospital Care System, Sarasota, Florida
  - Peoria Radiology Associates Research & Education Foundation, Peoria, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - St. Vincent Hospital & Health Care Center, Inc., Indianapolis, Indiana
  - The Care Group, LLC, Indianapolis, Indiana
  - Cardiovascular Institute of the South (CIS), Lafayette, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - NYPH & Trustees of Columbia University of New York, New York, New York
  - WakeMed, Raleigh, North Carolina
  - Philadelphia Health and Education Corp. d/b/a Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - North Central Heart Institute, Sioux Falls, South Dakota
  - St. Luke's Episcopal Hospital, Houston, Texas
  - CAMC Institute, Charleston, West Virginia

REFERENCES:
- [Result] Rocha-Singh K, Jaff MR, Lynne Kelley E; RENAISSANCE Trial Investigators. Renal artery stenting with noninvasive duplex ultrasound follow-up: 3-year results from the RENAISSANCE renal stent trial. Catheter Cardiovasc Interv. 2008 Nov 15;72(6):853-62. doi: 10.1002/ccd.21749. PMID 19006254